CLINICAL TRIAL: NCT02843113
Title: Stepping Up 4 Your Child: The Impact of an Educational Program and Social Case Work Involvement on Single Fathers
Brief Title: Stepping Up 4 Your Child
Acronym: 4yourchild
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Kentucky Cabinet for Health & Family Services (Unknown)
Responsible Party: Principal Investigator, Armon R. Perry, Associate Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15.1258
Record Dates: First submitted 2016-07-07; First posted 2016-07-25 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Parenting Education Curriculum; Parenting Education Curriculum + Case Management; Waiting List Control
Keywords: single father; parenting behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 4 Your Child Program (Experimental): Program integrates the provision of responsible parenting, economic stability, and relationship education services to fathers at risk for paternal disengagement.
  Interventions: Behavioral: 4 Your Child Program
- 4 Your Child + Case Management (Experimental): Participants assigned to treatment group that includes case management will receive an initial assessment to determine their strengths and needs. The participant will then work collaboratively with their case manager to connect to community resources to meet his needs. To do so, the case manager will meet with the participant using the following schedule: Months 1-2: intervention in the form of weekly face-to-face meeting with a case manager, plus a weekly phone call from a case manager; Months 3-4: intervention in the form of face-to-face meeting every other week, plus a weekly phone call; Months 5-6: intervention in the form of face-to-face meeting once a month, plus a weekly phone call.
  Interventions: Behavioral: 4 Your Child Program
- Waiting list control (No Intervention): Individuals who are randomly assigned to this condition will receive no treatment for a period of months in parallel with the experimental intervention conditions. Data will be gathered from them, and they will be randomly assigned to a treatment condition when possible.

INTERVENTIONS:
Behavioral: 4 Your Child Program — Integrates the provision of responsible parenting, economic stability, and relationship education services to fathers at risk for paternal disengagement.
  Arms: 4 Your Child + Case Management; 4 Your Child Program

SUMMARY:
Through Stepping Up 4 Your Child, non-custodial fathers will be provided with a comprehensive, solution-oriented program featuring group based parent education and individualized case management to help them achieve financial independence, increase their parenting skills, and develop a co-parenting alliance.

DETAILED DESCRIPTION:
Fathers' involvement in their children's lives has received increased attention in recent years. In response, support has grown for responsible fatherhood programs aimed at improving the quantity and quality of fathers' involvement. Research on these programs has concluded that factors such as fathers' parenting skills, co-parenting relationship quality, and socioeconomic status all impact fathers' ability to contribute to their children's growth and development. Using this previous research as a foundation, the Stepping Up 4 Your Child project will go beyond traditional fatherhood initiatives by integrating the provision of responsible parenting, economic stability, and relationship education services to fathers at risk for paternal disengagement. To do so, the University of Louisville's Kent School of Social Work will leverage its existing relationship with the Kentucky Office of Child Support Enforcement. Specifically, through Stepping Up 4 Your Child, non-custodial fathers will be provided with a comprehensive, solution-oriented program featuring group based parent education and individualized case management to help them achieve financial independence, increase their parenting skills, and develop a co-parenting alliance. Given that each of these focus areas have all been cited as three of the strongest predictors of paternal engagement, Stepping Up 4 Your Child and the results of its evaluation will have significant implications for the families it serves, as well as the practitioners, researchers, and policymakers interested in responsible fatherhood. 1

ELIGIBILITY:
Inclusion Criteria:

* non-custodial father AND
* age 16-24 OR
* age 24 up + low income OR
* age 24 up + child support payment delinquent

Exclusion Criteria:

* female
* custodial father
* male but not a father
* younger than age 16

Ages: 16 Years to 105 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1266 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Fathering Knowledge and Skills. | immediate after intervention, at 3 months later and at 6 months later
  Fathering knowledge and skills will be measured using the 24/7 Dad Fathering Skills Survey (National Fatherhood Initiative, 2010). This survey has 25 items that are multiple choice response questions. This survey comes with the 24/7 Dad curriculum packet. Given that this survey is a measure of fathering knowledge and not a standardized scale, no reliability data are available.
Change in Fathers' Parenting Behavior. | immediate after intervention, at 3 months later and at 6 months later
  Fathers' reported parenting behavior will be measured using the Index of Father Involvement (Hawkins et al., 2002). This measure has 9 factors loaded as subscales designed to tap direct and indirect forms of involvement and a total of 26 items. All items are measured on a 5 point scale ranging from A (excellent) to F (failing). The measure has a reported reliability/internal consistency score of .69
Change in Child Support Compliance. | immediate after intervention, at 3 months later and at 6 months later
  These payment data will be obtained via reports from the Kentucky Office of Child Support Enforcement.
Change in Co-Parenting Relationship Quality. | immediate after intervention, at 3 months later and at 6 months later
  Co-Parenting Relationship Quality. Co-parenting relationship quality will be measured using the Co-parenting Questionnaire (CQ, Margolis, Gordis, & John, 2001). This measure is a 14-item self-report instrument examining: 1) the amount of conflict between parents surrounding parenting issues, 2) cooperation as the extent to which mothers and fathers support, value, and respect each other as parents and the degree to which they ease one another's parenting burden, and 3) triangulation, the extent to which parents distort parent-child boundaries by attempting to form a coalition with the child that undermines or excludes the other parent. The 14 items form a three factor structure and have good internal consistency with alphas for the 3 factors and the total scale ranging from .69 to .87.

SECONDARY OUTCOMES:
Change in Conflict Resolution Skills. | immediate after intervention, at 3 months later and at 6 months later
  The Stanley-Markman Relationship Dynamics Scale (Renick et al, 1992) will be used to measure conflict resolution skills. This measure has reported Chronbach's alpha levels of .73 and .81 (Stanley et al, 2006) and strong predictive validity for relationship failure.
Change in Communication Skills. | immediate after intervention, at 3 months later and at 6 months later
  Communication skills will be measured through the Communication Patterns Questionnaire to assess communication skills. This measure has strong discriminant validity and Chronbach's alpha levels ranging from .73 to .88 (Noller & White, 1990).

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Elizabethtown, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Owensboro, Kentucky
  - Owenton, Kentucky
  - Paducah, Kentucky
  - Sandy Hook, Kentucky